CLINICAL TRIAL: NCT04302688
Title: Accurate Classification System for Patients With COVID-19 Based on Prognostic Nomogram
Brief Title: Accurate Classification System for Patients With COVID-19 Pneumonitis
Status: Completed | Type: Observational
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Principal Investigator, Gong Qiong, Professor, Renmin Hospital of Wuhan University
Other Study IDs: COVID-19 WU1
Record Dates: First submitted 2020-03-07; First posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Pneumonitis
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- modeling cohort: The 445 patients were grouped in chronological order.
- validating colort: The remaining 224 patients.

INTERVENTIONS:
Other:

SUMMARY:
The COVID-19 has a clustering morbidity trend and older people with chronic diseases are more likely to die, such as chronic renal insufficiency and chronic cardiovascular disease. We set up a COVID-19 pneumonia grading scale. The COVID-19 score system was validated to predict the clinical outcome of a patient.

DETAILED DESCRIPTION:
1. First we collect the medical records, according to the time sequence, the patients were divided into two groups, one is the model group, and the other is the validate group.
2. Responsible for the risk factor of regression equation according to the model. The patients were divided into three groups according to their total score of risk responsibility.
3. Compared with SEPSIS and CURB-65 grading system with the grading system we established.

ELIGIBILITY:
Inclusion Criteria:

* Patients with novel coronavirus pneumonia should be examined and diagnosed by CT and swab test of viral nucleic acid.

Exclusion Criteria:

* Patients who should have died during the course of the disease, but the cause of death was unrelated to viral pneumonia.
* Suspected patient review refers to the negative nucleic acid test.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with novel coronavirus pneumonia, and all cases were collected from the People's Hospital of Wuhan University.
Sampling Method: Non-Probability Sample
Enrollment: 669 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-03-04 (Actual)

PRIMARY OUTCOMES:
survival status | 10 December 2019 to 10 February 2020
  survival status as of February 24, 2020

CONTACTS AND LOCATIONS:
Overall Officials: Qiong Gong, MD., Principal Investigator — Renmin Hospital of Wuhan University
Locations (1):
- Renmin Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
Not going to share for the time being.